CLINICAL TRIAL: NCT04540224
Title: The Relationship Between the Differences in Blood Cytokine Values and Disease Stage in Luminal A, Luminal B and Triple Negative Breast Cancers.
Brief Title: The Relationship Between the Differences in Blood Cytokine Values in Breast Cancers.
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof. MD, Istanbul Training and Research Hospital
Other Study IDs: Breast Cancer
Record Dates: First submitted 2020-09-03; First posted 2020-09-07 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
Keywords: Luminal A; Luminal B; Triple Negative; Cytokine; Flow-Cytometry
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Luminal A: Breast cancer patients with Luminal A phenotype
  Interventions: Diagnostic Test: Flow-Cytometric analysis
- Luminal B: Breast cancer patients with Luminal B phenotype
  Interventions: Diagnostic Test: Flow-Cytometric analysis
- Triple Negative: Breast cancer patients with Triple negative phenotype
  Interventions: Diagnostic Test: Flow-Cytometric analysis
- Control: Healthy volunteers
  Interventions: Diagnostic Test: Flow-Cytometric analysis

INTERVENTIONS:
Diagnostic Test: Flow-Cytometric analysis — Measuring the level of serum IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1, IL-6, IL-8, IL-10, IL-12p (70), IL-17A, IL-18, IL-23 and IL-33

SUMMARY:
While classification of malignant breast tumors has traditionally been made according to their histological appearance, nowadays some subtypes have been defined according to their molecular features. The different behaviors of tumors in the luminal group necessitated the need to separate this group into luminal A and B subtypes. Luminal A group has the highest prevalence among breast cancers; It includes Her2 negative tumors with low proliferative activity, mitosis rate and low histological grade. The prognosis of patients with luminal A tumors is very good and metastases are often limited to bones. Luminal-B tumors are more aggressive. There are some studies investigating the relationship between blood cytokine levels (TGFβ1, IFNγ) and breast cancer. Human studies have generally evaluated a limited number of cytokines. The study evaluating the largest number of different cytokines was an animal study, and 24 different cytokine levels were compared with healthy control rats with breast cancer. Our aim in this study is to evaluate the relationship between the differences in blood cytokine values and disease stage in Luminal A, Luminal B, and triple negative breast cancers.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer in women and the second most common cause of death after lung cancer. In epidemiological studies, its prevalence is 22-26%, and the risk of mortality due to breast cancer is around 18%. While classification of malignant breast tumors has traditionally been made according to their histological appearance, nowadays some subtypes have been defined according to their molecular features. The different behaviors of tumors in the luminal group necessitated the need to separate this group into luminal A and B subtypes. Luminal A group has the highest prevalence among breast cancers; It includes Her2 negative tumors with low proliferative activity, mitosis rate and low histological grade. The prognosis of patients with luminal A tumors is very good and metastases are often limited to bones. Luminal-B tumors are more aggressive. The most important difference of this group is that tumors have a high proliferation rate. The breakpoint between Luminal A and B is generally accepted immunohistochemically as less than 14% of tumor cells show nuclear Ki67 expression. In addition, approximately 30% of Her2 positive tumors are immunohistochemically in the luminal B phenotype.

Infection and inflammation constitute approximately 25% of the causes of cancer.Cancers associated with inflammation usually occur as a result of mutations in DNA. Examples of cancers associated with chronic infections include Schistosoma haematobium-bladder cancer, Helicobacter pylori-stomach cancer, human papillomavirus-cervical cancer, Epstein-Barr virus-nasopharynx cancer, while chronic inflammation due to pro-inflammatory factors (asbestos, nanomaterials, Barrett's esophagus and ulcerative colitis etc.) plays a role in cancer development. Chronic inflammation also plays an important role in the development and recurrence of breast cancer. NF-κB pathway proteins, CRP, serum amyloid, matrix metalloproteinase enzyme family (MMP2, MMP9), urokinase type tissue plasminogen activators are associated with inflammatory cell migration and breast cancer.

There are some studies investigating the relationship between blood cytokine levels (TGFβ1, IFNγ) and breast cancer. Human studies have generally evaluated a limited number of cytokines. The study evaluating the largest number of different cytokines was an animal study, and 24 different cytokine levels were compared with healthy control rats with breast cancer.In this study we aimed to evaluate the relationship between the differences in blood cytokine values (IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1, IL-6, IL-8, IL-10, IL-12p (70), IL-17A, IL-18, IL-23 and IL-33) and disease stage in Luminal A, Luminal B, and triple negative breast cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer

Exclusion Criteria:

* Cancer Patients other than breast cancers
* Patients with known immunodeficiency
* Pregnancy
* Patients who had neoadjuvant chemoradiotherapy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — We want to evaluate the cytokine levels of female breast cancers
Study Population: In case group patients with breast cancers will be included to the study. Patients will be divided into subgroups according to the cancer receptor status.
  Also healty volunteers who don't have breast compliants will be the control group
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Serum cytokine levels | 6 months
  Serum Levels of serum IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1, IL-6, IL-8, IL-10, IL-12p (70), IL-17A, IL-18, IL-23 and IL-33

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Oguz Idiz, Assoc.Prof., Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murata M. Inflammation and cancer. Environ Health Prev Med. 2018 Oct 20;23(1):50. doi: 10.1186/s12199-018-0740-1. PMID 30340457
- [Background] Bera A, Russ E, Manoharan MS, Eidelman O, Eklund M, Hueman M, Pollard HB, Hu H, Shriver CD, Srivastava M. Proteomic Analysis of Inflammatory Biomarkers Associated With Breast Cancer Recurrence. Mil Med. 2020 Jan 7;185(Suppl 1):669-675. doi: 10.1093/milmed/usz254. PMID 32074342
- [Background] Vitiello GAF, Amarante MK, Oda JMM, Hirata BKB, de Oliveira CEC, Campos CZ, de Oliveira KB, Guembarovski RL, Watanabe MAE. Transforming growth factor beta 1 (TGFbeta1) plasmatic levels in breast cancer and neoplasia-free women: Association with patients' characteristics and TGFB1 haplotypes. Cytokine. 2020 Jun;130:155079. doi: 10.1016/j.cyto.2020.155079. Epub 2020 Mar 28. PMID 32229413